CLINICAL TRIAL: NCT00323492
Title: Open-label Randomized Multicenter Trial to Evaluate the Impact on the Lipid Profile of the Substitution of the NRTIs of a HAART Regimen by a Once Daily Fixed Dose Combination Tablet of Emtricitabine and Tenofovir DF Versus Maintained Treatment in HIV Infected Controlled Patients.
Brief Title: TOTEM: Switch From Other Nucleoside Reverse Transcriptase Inhibitors (NRTIs) to Once Daily Truvada
Acronym: TOTEM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Camille Aubron-Olivier, Gilead Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-FR-164-0109
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2009-12-23 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: HIV Infections
Keywords: HIV 1 Infection
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Truvada (Experimental): Truvada once daily with continuation of the current NNRTI or PI at randomization
  Interventions: Drug: Truvada
- Maintain Baseline Regimen (Active Comparator): Maintain baseline regimen
  Interventions: Drug: Current HAART regimen
- Delayed Truvada (Experimental): Truvada once daily with NNRTI or PI (participants from the comparator group who switched to Truvada during Study Phase 2)
  Interventions: Drug: Truvada
- All Truvada (Experimental): Truvada once daily with NNRTI or PI (all participants who received Truvada during the study, i.e., participants in the Truvada and Delayed Truvada groups)
  Interventions: Drug: Truvada

INTERVENTIONS:
Drug: Truvada — Truvada + NNRTI or PI.
  Arms: All Truvada; Delayed Truvada; Truvada
Drug: Current HAART regimen — Maintain baseline regimen
  Arms: Maintain Baseline Regimen

SUMMARY:
This study looked at lipid changes in human immunodeficiency virus type 1 (HIV-1) infected patients when the nucleoside reverse transcriptase inhibitors (NRTIs) in their existing highly active antiretroviral therapy (HAART) regimen were switched to Truvada® (a fixed dose combination tablet of emtricitabine/tenofovir disoproxil fumarate 200 mg/300 mg [FTC/TDF]). Subjects continued their nonnucleoside reverse transcriptase inhibitor (NNRTI) or protease inhibitor (PI) at the same dose.

DETAILED DESCRIPTION:
This was a Phase IV, multicenter (in France), open label study. The study was conducted in two phases: a comparative randomized phase, which served the primary objective of the study, and a follow-up phase.

Study Phase 1, Day -14 to Week 12: patients were randomized on a 1:1 basis to one of two groups:

* A. Truvada (substitution of their current NRTIs by Truvada [FTC/TDF] with continuation of their current NNRTI or PI at the same dose)
* B. Maintain Baseline Regimen (continuation of previous HAART regimen, i.e., maintained baseline regimen).

This phase of the study served the primary objective of the study.

Study Phase 2, roll-over follow-up, Week 12 to Week 48: Patients in the Truvada group continued with Truvada + an NNRTI or PI. Patients in the control group could switch their NRTIs to Truvada in this phase of the study (Delayed Truvada group).

Patients were assessed for efficacy and safety during both phases of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients displaying abnormal fasted triglycerides (> 2 g/L [2.26 mmol/L] and less than or equal to 10 g/L [11.29 mmol/L]) and/or fasted low density lipoprotein cholesterol (LDL-CHO; > 1.6 g/L [4.15 mmol/L])
* Patients on stable HAART with 2 NRTIs + 1 NNRTI or 1 PI for at least 3 months prior to screening, and with plasma viral load < 400 copies/mL for at least 6 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camille Aubron-Olivier, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Paris, France

REFERENCES:
- [Derived] Valantin MA, Bittar R, de Truchis P, Bollens D, Slama L, Giral P, Bonnefont-Rousselot D, Petour P, Aubron-Olivier C, Costagliola D, Katlama C; TOTEM trial group. Switching the nucleoside reverse transcriptase inhibitor backbone to tenofovir disoproxil fumarate + emtricitabine promptly improves triglycerides and low-density lipoprotein cholesterol in dyslipidaemic patients. J Antimicrob Chemother. 2010 Mar;65(3):556-61. doi: 10.1093/jac/dkp462. Epub 2010 Jan 6. PMID 20053692

RESULTS

PARTICIPANT FLOW:
Groups:
- Truvada: Truvada + nonnucleoside reverse transcriptase inhibitor (NNRTI) or protease inhibitor (PI).
- Delayed Truvada: Truvada + NNRTI or PI (participants from the control group who switched NRTIs to Truvada during Study Phase 2).
Period: Study Phase 1
Arm/Group | Truvada | Maintain Baseline Regimen | Delayed Truvada
Started | 47 | 45 | 0 (Not applicable to Phase 1.)
Intent-to-Treat (ITT) Analysis Set | 46 (One subject was excluded from ITT analysis set due to protocol violation.) | 45 | 0
Completed | 45 | 45 | 0
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Period: Study Phase 2
Arm/Group | Truvada | Maintain Baseline Regimen | Delayed Truvada
Started | 44 (1/45 subjects completed Phase 1 but did not start Phase 2. Week 48 ITT N=46) | 18 (2/45 subjects completed Phase 1 but did not start Phase 2. Week 48 ITT N=20 (no switch to Truvada)) | 25 (N=25 switched to Truvada in Phase 2.)
Completed | 40 | 17 | 24
Not Completed | 4 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Noncompliance with study schedule | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Truvada | Maintain Baseline Regimen | Total
Number analyzed (Participants) | 47 | 45 | 92
Age Continuous [Median (Inter-Quartile Range); unit: years] | 49.0 (10.7) [42.0 to 58.0] | 43.0 (7.7) [39.0 to 50.0] | 47.0 (9.8) [41.0 to 55.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 39 | 41 | 80
Region of Enrollment [Number; unit: participants]
  France | 47 | 45 | 92
Participants with plasma HIV-1 RNA < 400 copies/mL [Number; unit: participants] — At screening
  participants | 47 | 45 | 92
Cluster determinant 4 (CD4) cell count [Median (Inter-Quartile Range); unit: cells/mm^3] — At screening
  cells/mm^3 | 467 [314 to 698] | 559 [337 to 714] | 528 [318 to 709]
Low density lipoprotein cholesterol (LDL-CHO) [Median (Inter-Quartile Range); unit: mmol/L] — Centralized laboratory assessment
  mmol/L | 4.0 [3.2 to 4.7] | 4.0 [3.6 to 4.8] | 4.0 [3.4 to 4.7]
Triglycerides [Median (Inter-Quartile Range); unit: mmol/L] — Centralized laboratory assessment
  mmol/L | 2.3 [1.9 to 4.0] | 2.7 [1.9 to 3.6] | 2.4 [1.9 to 3.7]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Fasting Triglycerides
Description: Centralized laboratory assessment. Change = Week 12 value minus baseline value.
Time Frame: Baseline to Week 12
Population: ITT. Last post-baseline observation carried forward (LOCF) method was used for the analysis if the Week 12 value was missing. A missing datum were replaced by the last post-baseline value.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Truvada | Maintain Baseline Regimen
Number analyzed (Participants) | 44 | 45
mmol/L | -0.5 [-1.2 to 0.0] | -0.1 [-0.8 to 0.3]
Statistical Analysis 1: Comparison: Truvada vs Maintain Baseline Regimen; Null Hypothesis: changes from baseline in the two treatment groups are equal. Alternative Hypothesis: changes from baseline in the two treatment groups are different (two sided); Test type: Superiority or Other; p = 0.034, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were applied; Median Difference (Net) = -0.42, 95% CI [-0.86 to -0.03] — Difference is for Truvada minus Maintain Baseline Regimen. The non-parametric estimate of the difference between groups (Hodges-Lehmann) and its 95% confidence intervals (Moses) are provided

2. Primary Outcome: Change From Baseline to Week 12 in Fasting Low-density Lipoprotein Cholesterol (LDL-CHO)
Description: Centralized laboratory assessment. Change = Week 12 value minus baseline value.
Time Frame: Baseline to Week 12
Population: ITT. LOCF method was used for the analysis if the Week 12 value was missing. A missing datum were replaced by the last post-baseline value.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Truvada | Maintain Baseline Regimen
Number analyzed (Participants) | 44 | 45
mmol/L | -0.4 [-1.0 to 0.1] | -0.1 [-0.5 to 0.4]
Statistical Analysis 1: Comparison: Truvada vs Maintain Baseline Regimen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.031, Wilcoxon Rank Sum text — No adjustments for multiple comparisons were made; No adjustments were made; Median Difference (Net) = -0.36, 95% CI [-0.67 to -0.03] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline to Week 12 in Fasting High-density Lipoprotein Cholesterol (HDL-CHO)
Description: Centralized laboratory assessment. Change = Week 12 value minus baseline value.
Time Frame: Baseline to Week 12
Population: ITT. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Truvada | Maintain Baseline Regimen
Number analyzed (Participants) | 44 | 44
mmol/L | -0.1 [-0.2 to 0.1] | 0.0 [0.0 to 0.1]
Statistical Analysis 1: Comparison: Truvada vs Maintain Baseline Regimen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.009, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made; Median Difference (Net) = -0.10, 95% CI [-0.18 to -0.02] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline to Week 12 in Fasting Total Cholesterol (T-CHO)
Description: Centralized laboratory assessment. Change = Week 12 value minus baseline value.
Time Frame: Baseline to Week 12
Population: ITT. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Truvada | Maintain Baseline Regimen
Number analyzed (Participants) | 44 | 44
mmol/L | -0.8 [-1.3 to -0.1] | -0.1 [-0.7 to 0.5]
Statistical Analysis 1: Comparison: Truvada vs Maintain Baseline Regimen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Wicoxon Rank Sum test — No adjustments for multiple comparisons were made; no adjustments were made; Median Difference (Net) = -0.64, 95% CI [-1.01 to -0.27] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline to Week 12 in Fasting T-CHO/HDL-CHO
Description: Centralized laboratory assessment. Change = Week 12 value minus baseline value.
Time Frame: Baseline to Week 12
Population: ITT. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Truvada | Maintain Baseline Regimen
Number analyzed (Participants) | 44 | 44
Ratio | -0.5 [-0.7 to 0.2] | -0.1 [-0.8 to 0.3]
Statistical Analysis 1: Comparison: Truvada vs Maintain Baseline Regimen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.51, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made; Median Difference (Net) = -0.10, 95% CI [-0.44 to 0.19] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline to Week 12 in Fasting HDL-CHO/LDL-CHO
Description: Centralized laboratory assessment. Change = Week 12 value minus baseline value.
Time Frame: Baseline to Week 12
Population: ITT. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Truvada | Maintain Baseline Regimen
Number analyzed (Participants) | 44 | 44
Ratio | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.1]
Statistical Analysis 1: Comparison: Truvada vs Maintain Baseline Regimen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.79, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made; Median Difference (Net) = 0.0, 95% CI [-0.03 to 0.02] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline to Week 12 in Fasting Ultra-sensitive C-reactive Protein (Us-CRP)
Description: Local laboratory assessment. Change = Week 12 value minus baseline value.
Time Frame: Baseline to Week 12
Population: ITT. Missing values were excluded. Assessment of us-CRP was added to the study schedule via protocol amendment part way through the study. This resulted in small numbers of subjects having data available for this analysis.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Truvada | Maintain Baseline Regimen
Number analyzed (Participants) | 16 | 7
mg/L | 0.4 [-0.5 to 0.9] | 0.7 [-3.2 to 2.5]
Statistical Analysis 1: Comparison: Truvada vs Maintain Baseline Regimen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.86, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

8. Secondary Outcome: Percentage of Participants With Fasting Plasma Triglycerides > 10 g/L (> 11.29 mmol/L) at Week 12
Description: Centralized laboratory assessment
Time Frame: 12 weeks
Population: ITT. Missing values were excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | Truvada | Maintain Baseline Regimen
Number analyzed (Participants) | 44 | 44
Percentage of participants | 0 | 0

9. Secondary Outcome: Change From Baseline to Week 12 in Cluster Determinant 4 (CD4) Cell Count
Description: Change = Week 12 value minus baseline value.
Time Frame: Baseline to Week 12
Population: ITT. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Truvada | Maintain Baseline Regimen
Number analyzed (Participants) | 44 | 44
cells/mm^3 | 17.5 [-36.0 to 63.5] | 16.0 [-31.0 to 92.0]
Statistical Analysis 1: Comparison: Truvada vs Maintain Baseline Regimen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.65, Wilcoxon Rank Sum test — No adjustments for multiple comparisons were made; No adjustments were made

10. Secondary Outcome: Change From Baseline to Week 48 in CD4 Cell Count
Description: Change = Week 48 value minus baseline value.
Time Frame: Baseline to Week 48
Population: ITT. Missing values were excluded.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Truvada | Maintain Baseline Regimen
Number analyzed (Participants) | 39 | 16
cells/mm^3 | 35.0 [-37.0 to 116.0] | 40.0 [-41.5 to 79.5]
Statistical Analysis 1: Comparison: Truvada; Null Hypothesis: no indication of shift from 0 in distribution of change from baseline. Alternative Hypothesis: shift from 0 is observed in distribution of change from baseline; Test type: Superiority or Other; p = 0.11, Wilcoxon Signed Rank test — No adjustments were made; No adjustments were made
Statistical Analysis 2: Comparison: Maintain Baseline Regimen; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.34, Wilcoxon Signed Rank test — No adjustments were made; No adjustments were made

11. Secondary Outcome: Percentage of Participants With Virologic Control (Plasma HIV-1 Ribonucleic Acid [RNA] < 400 Copies/mL) at Week 12
Time Frame: 12 weeks
Population: ITT. Missing values were treated as failure.
Measure: Number; unit: Percentage of participants
Arm/Group | Truvada | Maintain Baseline Regimen
Number analyzed (Participants) | 46 | 45
Percentage of participants | 96 | 98
Statistical Analysis 1: Comparison: Truvada vs Maintain Baseline Regimen; Null Hypothesis: treatment is not associated with the observed virologic response. Alternative Hypothesis: treatment is associated with the observed virologic response; Test type: Superiority or Other; p = 1.00, Fisher Exact — No adjustments were made; No adjustments were made

12. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Greater Than or Equal to 400 Copies/mL at Week 12
Time Frame: 12 weeks
Population: ITT. Missing values were excluded. Any subjects with plasma HIV-1 RNA greater than or equal to 400 copies/mL at Week 12 were to have virologic genotyping performed.
Measure: Number; unit: Percentage of participants
Arm/Group | Truvada | Maintain Baseline Regimen
Number analyzed (Participants) | 46 | 45
Percentage of participants | 0 | 0

13. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA < 400 Copies/mL at Week 48
Time Frame: 48 weeks
Population: ITT. Missing values were treated as failure.
Measure: Number; unit: Percentage of participants
Arm/Group | Truvada | Maintain Baseline Regimen
Number analyzed (Participants) | 46 | 20
Percentage of participants | 80 | 80

ADVERSE EVENTS:
Groups:
- Truvada: Truvada + NNRTI or PI. The number of participants at risk is the number who started the study by switching to Truvada. Participants in this group were to remain on Truvada for 48 weeks (duration of the study). The number at risk was reduced only by study discontinuation (from 47 at baseline to 40 who completed Study Phase 2).
- Maintain Baseline Regimen: Maintain baseline regimen. The number of participants at risk is the number who started the study by maintaining their baseline regimen. Per protocol, participants in this group were allowed to switch to Truvada after Week 12 (Delayed TVD group), therefore the number of participants at risk declines over time (from 45 at baseline to 17 who completed Study Phase 2; with most participants switching to Truvada at Week 12).
- All Truvada: Truvada + NNRTI or PI (all participants who received Truvada during the study, i.e., participants in the Truvada and Delayed Truvada groups). The number of participants at risk is the number who started the study by switching to Truvada (Truvada group), plus those who started the study by maintaining their baseline regimen but who switched to Truvada during the study (Delayed Truvada group). The number of participants at risk increases over time (from 47 at baseline to 72 when the last switch to Truvada took place; 25 participants switched to Truvada from the "maintain baseline regimen" group in Study Phase 2).
Arm/Group | Truvada | Maintain Baseline Regimen | All Truvada
Serious Adverse Events (participants affected / at risk) | 7/47 | 3/45 | 7/72
Other Adverse Events (participants affected / at risk) | 15/47 | 6/45 | 16/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Truvada (N=47) | Maintain Baseline Regimen (N=45) | All Truvada (N=72)
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0 | 2
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Truvada (N=47) | Maintain Baseline Regimen (N=45) | All Truvada (N=72)
Bronchitis (Infections and infestations) | 3 | 2 | 3
Herpes simplex (Infections and infestations) | 3 | 0 | 3
Nasopharyngitis (Infections and infestations) | 3 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 7
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Pollakiuria (Renal and urinary disorders) | 3 | 0 | 3

LIMITATIONS AND CAVEATS:
Comparison of adverse events between Truvada and maintain baseline regimen groups is inappropriate since numbers at risk (and exposure to study drug) are not balanced, as described in the adverse event treatment group descriptions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead Sciences, investigators in this study may communicate, orally present, or publish in scientific journals or other scholarly media only after the following conditions have been met: results of the study in their entirety have been publicly disclosed by or with the consent of Gilead Sciences in an abstract, manuscript, or presentation form; or study has been completed at all study sites for at least 2 years.